CLINICAL TRIAL: NCT03341559
Title: Spatial Frequency Domain Imaging (SFD) for Assessment of Diabetic Foot Ulcer Development and Healing
Status: Completed | Type: Observational
Sponsor: University of Southern California (Other)
Collaborators: Modulated Imaging Inc. (Industry)
Responsible Party: Principal Investigator, David Armstrong, Professor of Surgery and Director, Southwestern Academic Limb Salvage Alliance (SALSA), University of Southern California
Other Study IDs: APP-17-06886
Record Dates: First submitted 2017-11-06; First posted 2017-11-14 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

GROUPS / COHORTS (2):
- With Existing Diabetic Ulcers: Current DFU
  Interventions: Device: Spatial Frequency Domain Imaging (SFDI)
- Diabetic Ulcers in remission: DFU in remission
  Interventions: Device: Spatial Frequency Domain Imaging (SFDI)

INTERVENTIONS:
Device: Spatial Frequency Domain Imaging (SFDI) — Observational study to measure perfusion in lower extremities for prediction of both healing and formation of diabetic foot ulcers using Reflect RS
  Other Names: Reflect RS

SUMMARY:
This study is designed to evaluate the ability of Spatial Frequency Domain Imaging (SFDI) to measure perfusion in lower extremities for prediction of both healing and formation of diabetic foot ulcers.

The investigators will perform longitudinal imaging (for 12 months) in two cohorts of subjects

ELIGIBILITY:
Inclusion Criteria:

I. Will be followed up in clinic on monthly basis for the next 12 months per standard of care II. Belong to one of the two target groups

1. Subjects with an existing diabetic foot ulcer
2. Subjects determined "at risk" for an ulcer

Exclusion Criteria:

1. History of heart failure
2. Rheumatoid arthritis
3. Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male or female patients at University of Southern California diagnosed with a Diabetic Foot Ulcer
Sampling Method: Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2018-03-20 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-02-13 (Actual)

PRIMARY OUTCOMES:
Perfusion in lower extremities | 12-month
  SFDI data outputs

CONTACTS AND LOCATIONS:
Locations (1):
- Keck Medical Center of USC, Los Angeles, California, United States

REFERENCES:
- [Derived] Murphy GA, Singh-Moon RP, Mazhar A, Cuccia DJ, Rowe VL, Armstrong DG. Quantifying dermal microcirculatory changes of neuropathic and neuroischemic diabetic foot ulcers using spatial frequency domain imaging: a shade of things to come? BMJ Open Diabetes Res Care. 2020 Nov;8(2):e001815. doi: 10.1136/bmjdrc-2020-001815. PMID 33219118